CLINICAL TRIAL: NCT05592860
Title: Comparison of Glycemic Control With Smartphone Application (Vivovitals) - Based Glucose Monitoring to Routine Home Glucose Monitoring in Poorly Controlled T2DM Patients Treated With Insulin
Brief Title: Comparison of Glycemic Control With Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Issac Sachmechi, Director of Diabetes Center of Excellence, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-20-01694; FWA#00005656 (Other: Department of Health and Human Services); FWA#00005651 (Other: Department of Health and Human Services)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile application (Experimental): Mobile application to enter glucose level
  Interventions: Device: Mobile application
- Daily Diary (Placebo Comparator): Daily Diary to record glucose level
  Interventions: Behavioral: Daily Diary

INTERVENTIONS:
Device: Mobile application — participants in intervention group will use smart phone application and update glucose level and investigator will adjust the insulin accordingly
  Other Names: device related insulin adjustment
  Arms: Mobile application
Behavioral: Daily Diary — participants will use daily diary to record glucose level
  Arms: Daily Diary

SUMMARY:
The study is aimed to determine if a smartphone application based weekly glucose monitoring by a care provider is superior to the routine home glucose monitoring by patients in poorly controlled type 2 diabetes mellitus who are on insulin.

DETAILED DESCRIPTION:
The study is a randomized, prospective cohort study. Subjects will be enrolled randomly after fulfilling the meeting criteria into two groups. Group 1 (intervention group) will used mobile application to enter their glucose level and group 2 (control group) will record their glucose level on daily diary. Data collection will be standardized in order to eliminate bias. In addition, all statistical analyses will be performed by a departmental statistician and not the study investigators. Patients in each arm of the study will be selected form the same population in order to avoid selection bias.

ELIGIBILITY:
Inclusion Criteria:

* Adult type 2 diabetes mellitus patients (≥ 18years of age) whose HbA1c is ≥8% on insulin.
* At least three months of daily home glucose monitoring before including in the study
* Willing to provide consent to participate in the study4. Uses a smartphone with cellular network and willing to and has ability to learn and use the Vivo vitals application on it.

Exclusion Criteria:

* Patients who have Gestational diabetes or type 1 diabetes
* Patients who have been admitted to the hospital in the last month for more than 3 days.
* Patients who have adrenal disorders or taking exogenous glucocorticoids.
* Patients who are mentally incompetent, having uncontrolled psychiatric conditions, inmates.
* Patients with active malignancies including those on treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | at the end of 3 months follow-up
  A1C is a lab test that shows the average level of blood sugar (glucose) over the previous 3 months. It shows how well a person is controlling their blood sugar to help prevent complications from diabetes.

SECONDARY OUTCOMES:
Change in weight | baseline and 3 month
  Change in weight
Change in Body Mass Index (BMI) | baseline and 3 month
  Change in BMI
Change in blood pressure | baseline and 3 month
  Change in blood pressure - systolic and diastolic

CONTACTS AND LOCATIONS:
Overall Officials: Issac sachmechi, MD, FACE, FACP, Principal Investigator — Icahn school of medicine Mount Sinai
Locations (1):
- Queens Hospital Center, Jamaica, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee) identified for this purpose. To achieve aims in the approved proposal. Proposals should be directed to sachmeci@nychhc.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.

DOCUMENTS (1):
  • Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT05592860/ICF_000.pdf